CLINICAL TRIAL: NCT04283812
Title: A Re-attachable Stereotactic Frame System for Clinical Interventive Neurosurgery
Brief Title: New Stereotactic Frame System for Neurosurgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Per PI discretion, study closed and no participants enrolled
Sponsor: Mayo Clinic (Other)
Collaborators: NaviNetics Inc. (Unknown)
Responsible Party: Principal Investigator, Kai J. Miller, Principle Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 18-011914
Record Dates: First submitted 2020-02-23; First posted 2020-02-25 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Parkinson Disease; Essential Tremor; Dystonia; Tourette Syndrome; Obsessive-Compulsive Disorder
Keywords: deep brain stimulation; sterotactic surgery; neurological disorders; stereotactic instruments
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia; Tourette Syndrome; Obsessive-Compulsive Disorder; Nervous System Diseases

STUDY DESIGN:
Masking Description: No other parties will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- D1 Stereotactic System Assessment (Experimental): Participants in the clinical study will consist of subjects approved to undergo deep brain stimulation surgery for the treatment of a neurological disorder at Mayo Clinic. Subjects will have a Key secured to their skull for attachment of an MRI-compatible localizer box or D1 stereotactic frame. 3D Euclidian distance error(s), trajectory accuracy(s), operating room time, and comfort level of the system will be assessed.
  Interventions: Device: DBS Electrode Implantation using D1 Sterotactic System

INTERVENTIONS:
Device: DBS Electrode Implantation using D1 Sterotactic System — Treatment intervention will consist of subjects undergoing Mayo Clinic standard deep brain stimulation surgery specific to their diagnosed neurological disorder consisting of implantation of stimulating electrodes using the D1 stereotactic system.

SUMMARY:
This study is designed to demonstrate an in-house developed re-attachable stereotactic system that can markedly reduce the overall deep brain stimulation (DBS) procedure time to greatly facilitate subject access to neurosurgical restorative therapies. Subjects will consist exclusively of individuals who have been approved to undergo deep brain stimulation surgery for the treatment of a neurological disorder at Mayo Clinic - Rochester MN. This study is a quantitative comparative, between-subject study enrolling approximately 10 subjects.

DETAILED DESCRIPTION:
Aims:

This study will evaluate a new stereotactic device (D1 stereotactic system) designed to address shortcomings of current stereotactic systems by using a novel surface-mounted stereotactic system that is comparatively small, lightweight, user-friendly, and comparable in precision and accuracy to current clinical systems.

Methods:

Subjects will be recruited exclusively from adult subjects with a neurological disease. These subjects will be identified preoperatively from DBS clinical subjects. Each subject will undergo an evaluation by the Mayo Clinic Deep Brain Stimulation Committee (comprised of neurologists, neuropsychologists, psychiatrists, neurosurgeons, and radiologists) to receive a DBS surgery at Mayo Clinic - Rochester for the treatment of a neurological disease. All subjects will be pre-screened against the standard Mayo Clinic inclusion/exclusion criteria for DBS surgery through face-to-face interviews. Once a subject has been identified, the Study Coordinator will contact the subject for interest in participation in the study.

Step-by-Step Schedule:

Skull Anchor Key Attachment Location: St. Mary Hospital - Subject Preparation Room

1. Superior portion of the head, the hair is clipped off in the area where Skull Anchor Key would be placed. The clipped area and surrounding region is prepped in usual sterile fashion. This begins subject participation in the protocol.
2. The MR Localizer Box is placed upside down and the Skull Anchor Key is placed within its slot in the MR Localizer Box and screwed in using MR compatible screws.
3. The apparatus is positioned on the subject head and allowed to rest such that the Skull Anchor Key is midline and the ear bars lie parallel to the external auditory meatus taking caution to prevent the bottom surface of the Skull Anchor Key or the safety caps from becoming non sterile.
4. The Z value of the ear bars is adjusted such that the ear probes are at same horizontal level as the external auditory meatus. The ear bars are gently pushed into the external auditory meatus on both sides such that it is snug but comfortable to the subject. (NOTE: If required, the Y position of the ear bars may be readjusted at this step in situations such as the anterior N fiducial bars hitting the forehead of the subject).
5. After confirming accurate initial placement of the MR Localizer Box, the sites of skull screw and pins placement are marked using a surgical pen with the guide Skull Anchor Key which has holes instead of screws and pins acting as reference guide. The MR Localizer Box is then removed and each of the pen marked site receives an injection of local anesthetic.
6. Following local anesthetic application, the ear bars are removed from the ear while an assistant supports the MR Localizer Box. The MR Localizer Box is gradually lowered to allow the pins to penetrate scalp until it rests on the bone. At this point, titanium self-tapping screws are gently screwed in through the hole on each of the 2 angled legs of the Skull Anchor Key until the Skull Anchor Key is level and secure.
7. The subject is then transferred to the MR/CT Imaging Facility for target planning.

MRI Acquisition and Target Planning Location: St. Mary Hospital - Neuroradiology Facility

1. Once in MR suite, the subject rests their head in a custom made MR headrest which sits within the lower portion of RF coil. The headrest holds the axis of MR Localizer Box parallel to the axis of MR gantry and allows the frame to be held securely during the MR imaging.
2. The subject is positioned in a MR scanner in a supine position.
3. An anatomical image volume is acquired. The field of view region is adjusted to ensure the MR Localizer Box fiducials are visible in the MR images and then all images are acquired.
4. The images are then transferred to the surgical planning computer.
5. Following image acquisition, the images are reviewed by the surgical team to judge whether they are suitable for surgical planning. (If found unsuitable, the imaging and review is repeated.) Once satisfactory images are obtained, the subject is moved to the subject preparation room where the MR Localizer Box is detached from the KEY.
6. A DBS surgical plan, comprised of the electrode stereotactic target coordinates and an optimal trajectory is created by the navigational software. The plan is documented and shared with the surgical team.
7. The subject is then transferred to the operating room for DBS electrode implantation.

DBS Electrode Implantation Location: St. Mary Hospital - Operating Room

1. The subject is shifted to the operating room.
2. The D1 stereotactic device is attached to the Skull Anchor Key and the X, Y, Z, Arc and Collar angles will be adjusted based on MR planned coordinates.
3. Standard procedure is followed for making the incision and burr hole, putting in the DBS electrode, electrophysiologic target confirmation (as required) and securing the electrode in place.
4. A C-arm is then used to obtain a lateral view radiograph to confirm correct placement of the DBS electrode as assessed by the alignment of the tip of the DBS electrode with X-ray reticules on the stereotactic device.
5. Above steps are repeated for additional DBS electrode insertion.
6. After securing the last DBS electrode the stereotactic device is removed from the KEY. All DBS electrodes are then coiled and secured under the skin or are tunneled beneath the skin of the scalp and neck for battery placement as currently practiced. All surgical incisions are then sutured.
7. The CT Localizer Box is attached to the Skull Anchor Key to acquire a post-operative CT scan.
8. The subject is then transferred to the Neuroradiology Facility for post-operative CT imaging.

CT Confirmation and CT Localizer Box and KEY Removal Location: St. Mary Hospital - Neuroradiology Facility

1. With the subject in the CT imaging room the subject is positioned supine in the CT scanner to acquire a postoperative anatomical image volume to confirm the placement of the DBS electrode placement using planning software normally used for neurosurgical procedures.
2. Immediately following the CT scan, the subject is taken to the preparation room for removal of the CT Localizer Box, the Skull Anchor Key, and post-removal treatments. The self-tapping titanium screws are removed and the surgical site is treated appropriately.

Power Statement:

This is a pilot study with a unique subject cohort.

Data Analysis Plan:

The effectiveness of the D1 Stereotactic System in accurately implanting DBS electrodes in adults approved for DBS surgery at Mayo Clinic for treatment of a neurological disease will be evaluated by analyzing the following:

1. A 3D Euclidian distance error between the MR planned coordinate (XP, YP, ZP) and CT confirmed actual DBS coordinate (XA, YA, ZA) will be calculated. The 3D distance error comparable or lower to conventional system will be accounted as success criteria. Unpaired t-test will be used to determine whether the difference is significantly different or not.
2. A trajectory accuracy will be determined by comparing Collar Angle (CA) and Arc Angle (AA) between MR planned angles (CAP and AAP) and CT confirmed actual angles (CAA and AAA). The non-significant difference between MR planned and CT confirmed angles will be accounted as success criteria. Paired t-test will be used for 10 patient data.
3. Operating room time will be counted and compared to conventional procedure (using Leksell frame). The average operating room time will be compared between conventional procedure and D1 Stereotactic System procedure. Significantly lower operating room time will be accounted as success criteria.
4. Comfort level questionnaire will be given to each subject after DBS surgery and removal of the device to assess their overall experience with device and surgery.

Data Exclusion Criteria: If any surgical plan is changed in operating room (i.e., target coordinate, trajectory), the data will be excluded. However, the change of DBS electrode depth will be accounted as valid data.

ELIGIBILITY:
Inclusion Criteria:

* Must be adult subjects with medically intractable neurological disorder who have been approved for DBS surgery by the interdisciplinary Mayo DBS committee.
* Competent and willing to provide signed, informed consent to participate in the study.
* Competent and willing to provide written, informed consent to participate in the study.

Exclusion Criteria:

* Pregnant subjects, prisoners, individuals ages less than 18 and any subjects identified as unsuitable for DBS surgery by the Mayo Clinic DBS committee.
* Subjects unable to communicate with the investigator and staff.
* Any health condition that in the investigator's opinion should preclude participation in this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
3D Euclidian distance error | Within 1 month post-DBS surgery.
  3D Euclidian distance error between the MR planned coordinate (XP, YP, ZP) and CT confirmed actual DBS coordinate (XA, YA, ZA) will be calculated. The 3D distance error comparable or lower to conventional system will be accounted as success criteria.
Trajectory accuracy | Within 1 month post-DBS surgery.
  A trajectory accuracy will be determined by comparing Collar Angle (CA) and Arc Angle (AA) between MR planned angles (CAP and AAP) and CT confirmed actual angles (CAA and AAA). The non-significant difference between MR planned and CT confirmed angles will be accounted as success criteria.
Operating room time | Within 1 month post-DBS surgery.
  Operating room time will be counted and compared to conventional procedure (using Leksell frame). The average operating room time will be compared between conventional procedure and D1 Stereotactic System procedure. Significantly lower operating room time will be accounted as success criteria
Comfort level questionnaire | Within 1 month post-DBS surgery.
  Comfort level questionnaire will be given to each subject after DBS surgery and removal of the device to assess their overall experience with device and surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Miller, MD, PhD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ben-Haim S, Falowski SM. Evaluation of Patient Perspectives Toward Awake, Frame-Based Deep-Brain Stimulation Surgery. World Neurosurg. 2018 Mar;111:e601-e607. doi: 10.1016/j.wneu.2017.12.122. Epub 2017 Dec 28. PMID 29288853
- [Background] Bjartmarz H, Rehncrona S. Comparison of accuracy and precision between frame-based and frameless stereotactic navigation for deep brain stimulation electrode implantation. Stereotact Funct Neurosurg. 2007;85(5):235-42. doi: 10.1159/000103262. Epub 2007 May 25. PMID 17534136
- [Background] Bot M, van den Munckhof P, Bakay R, Sierens D, Stebbins G, Verhagen Metman L. Analysis of Stereotactic Accuracy in Patients Undergoing Deep Brain Stimulation Using Nexframe and the Leksell Frame. Stereotact Funct Neurosurg. 2015;93(5):316-25. doi: 10.1159/000375178. Epub 2015 Jul 29. PMID 26227179
- [Background] Edwards CA, Rusheen AE, Oh Y, Paek SB, Jacobs J, Lee KH, Dennis KD, Bennet KE, Kouzani AZ, Lee KH, Goerss SJ. A novel re-attachable stereotactic frame for MRI-guided neuronavigation and its validation in a large animal and human cadaver model. J Neural Eng. 2018 Dec;15(6):066003. doi: 10.1088/1741-2552/aadb49. Epub 2018 Aug 20. PMID 30124202
- [Background] Goerss S, Kelly PJ, Kall B, Alker GJ Jr. A computed tomographic stereotactic adaptation system. Neurosurgery. 1982 Mar;10(3):375-9. doi: 10.1227/00006123-198203000-00014. PMID 7041006
- [Background] Grahn PJ, Goerss SJ, Lujan JL, Mallory GW, Kall BA, Mendez AA, Trevathan JK, Felmlee JP, Bennet KE, Lee KH. MRI-Guided Stereotactic System for Delivery of Intraspinal Microstimulation. Spine (Phila Pa 1976). 2016 Jul 1;41(13):E806-E813. doi: 10.1097/BRS.0000000000001397. PMID 26679880
- [Background] Kelly PJ, Kall BA, Goerss S. Computer simulation for the stereotactic placement of interstitial radionuclide sources into computed tomography-defined tumor volumes. Neurosurgery. 1984 Apr;14(4):442-8. doi: 10.1227/00006123-198404000-00009. PMID 6374493
- [Background] Kelly PJ, Sharbrough FW, Kall BA, Goerss SJ. Magnetic resonance imaging-based computer-assisted stereotactic resection of the hippocampus and amygdala in patients with temporal lobe epilepsy. Mayo Clin Proc. 1987 Feb;62(2):103-8. doi: 10.1016/s0025-6196(12)61877-1. PMID 3543519
- [Background] Knight EJ, Min HK, Hwang SC, Marsh MP, Paek S, Kim I, Felmlee JP, Abulseoud OA, Bennet KE, Frye MA, Lee KH. Nucleus accumbens deep brain stimulation results in insula and prefrontal activation: a large animal FMRI study. PLoS One. 2013;8(2):e56640. doi: 10.1371/journal.pone.0056640. Epub 2013 Feb 18. PMID 23441210
- [Background] Konrad PE, Neimat JS, Yu H, Kao CC, Remple MS, D'Haese PF, Dawant BM. Customized, miniature rapid-prototype stereotactic frames for use in deep brain stimulator surgery: initial clinical methodology and experience from 263 patients from 2002 to 2008. Stereotact Funct Neurosurg. 2011;89(1):34-41. doi: 10.1159/000322276. Epub 2010 Dec 15. PMID 21160241
- [Background] Min HK, Ross EK, Lee KH, Dennis K, Han SR, Jeong JH, Marsh MP, Striemer B, Felmlee JP, Lujan JL, Goerss S, Duffy PS, Blaha C, Chang SY, Bennet KE. Subthalamic nucleus deep brain stimulation induces motor network BOLD activation: use of a high precision MRI guided stereotactic system for nonhuman primates. Brain Stimul. 2014 Jul-Aug;7(4):603-607. doi: 10.1016/j.brs.2014.04.007. Epub 2014 May 2. PMID 24933029
- [Background] Okun MS, Fernandez HH, Rodriguez RL, Foote KD. Identifying candidates for deep brain stimulation in Parkinson's disease: the role of the primary care physician. Geriatrics. 2007 May;62(5):18-24. PMID 17489644
- [Background] Wang DD, Lau D, Rolston JD, Englot DJ, Sneed PK, McDermott MW. Pain experience using conventional versus angled anterior posts during stereotactic head frame placement for radiosurgery. J Clin Neurosci. 2014 Sep;21(9):1538-42. doi: 10.1016/j.jocn.2014.02.009. Epub 2014 May 6. PMID 24814855
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials